CLINICAL TRIAL: NCT05957627
Title: Effect of Saleem's Protocol on Foot Deformity in Congenital Talipes Equinovarus
Brief Title: Management of Congenital Talipes Equinovarus by Saleem's Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Society for Rehabilitation of Differently Abled Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSRD Hospital
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Congenital Talipes Equinovarus
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Saleem's intervention (Experimental): Early tenotomies and serial casting were used in Saleem's technique to reduce foot deforming forces. It involved 2 principal tenotmies and 2 accessory tenotmies. Principal tenotmies include tendo achillies and planter fascia release. 2 Accessory tenotmies include tibialis posterior and abductor hallucis. All tenotmies are done under local anesthesia.The foot is placed in a serial cast close to its natural anatomical position following tenotomies at first visit. children are evaluated after 1 week.This technique necessitates 4 to 5 casts on average. DB shoes were advised when the foot casting was finished, and a 6-month follow-up with the patient was conducted.
  Interventions: Procedure: Saleem's protocol

INTERVENTIONS:
Procedure: Saleem's protocol — It involved 2 principal tenotmies and 2 accessory tenotmies. Principal tenotmies include tendo achillies and planter fascia release. 2 Accessory tenotmies include tibialis posterior and abductor hallucis. All tenotmies are done under local anesthesia

SUMMARY:
The main objective of this study is to evaluate the effectiveness of Saleem's protocol treatment plan for congenital ideopathic talipes equino varus deformity using early tenotomy and serial foot casting. The combined effect of early tenotomies and foot serial casting has not been proven in prior investigations. Ten kids were involved in this pilot study where Saleem's protocol approach was used. With the use of the PIRANI score, the baseline reading was evaluated. Readings were obtained before each cast performance. This study results show's early correction of foot deformity with average 4 to 5 cast and no recurrence.

DETAILED DESCRIPTION:
Congenital idiopathic clubfoot, also known as congenital talipes equinovarus, is the most common serious musculoskeletal birth defect that occurs in the United States and the world. Idiopathic clubfoot occurs in otherwise normal infants and should be distinguished from syndromic clubfoot and neurogenic clubfoot, which occur in infants as part of a syndrome or neurologic condition.Clubfoot is one of the most common congenital abnormalities affecting the lower limb, it remains a challenge not only to understand its genetic origins but also to provide effective long-term treatment. Various environmental influences have been shown to increase the risk of clubfoot in that they may affect the developing foetus in different ways including via genetic alterations, deformation, or growth arrest. The incidence has been reported to rise with increased maternal alcohol consumption], smoking, and if the mothers had undergone amniocentesis especially where a leak of amniotic fluid had occurred. In a clubfoot the soft tissues are more resistant to pressure than the bones.Untreated clubfoot causes life-long impairment, affecting individuals' ability to walk and participate in society.It can be isolated or associated with other serious congenital abnormalities, especially if bilateral and severe. The ideal aim of treatment is to achieve a functional, pain-free, plantigrade foot in the long term. Pirani scoring system is one of the classification systems and is simple, easy to use in the management of clubfoot.The Pirani scoring system works by assessing six clinical signs of contracture, which may score 0 (no deformity), 0.5 (moderate deformity) or 1(severe deformity). The total score is recorded after every visit. Pirani scoring is known to be valid and reliable for providing a good forecast about the potential treatment for an individual foot, such that a higher score at presentation may indicate the requirement of a higher number of casts to correct the deformity.

Different types of conservative methods (Ponseti techniques, Kite's method, and French physical therapy method). Six to 12 numbers of casts (mean: 10) were required in ponseti method to obtain correction of clubfoot deformities. Mean period of immobilization in a cast was 13.9 weeks (10-15 weeks). However, relapses are common in severe clubfeet and are probably caused by the same pathology that initiated the deformity. The rate of recurrence after using the Ponseti method, occurring in up to 40% of patient.Compliance with the Ponseti protocol is a major problem and has a direct effect on the success of treatment. Numerous surgeons have performed complete, plantar, lateral, medial, and posterior releases with poor results.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital idiopathic clubfoot
* Both male and female under 1 year of age
* Participiants who are willing to participate

Exclusion Criteria:

* Childrens who suffer from neuropathy
* Childrens with syndromic club foot
* Childrens have done ponsetti before
* Childrens with foot drop
* Above 1 year of age

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-08-25 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
PIRANI Score | 6 months
  The Pirani Score is a simple and reliable system to determine severity and monitor progress in the Assessment and Treatment of Clubfoot.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Saleem Bashir, FCPS, Study Director — Pakistan Society for Rehabilitation of Differently Abled Hospital; Nayab Iqbal, MS, Principal Investigator — PSRD
Locations (1):
- Pakistan Society for the Rehabilitation of Diffrently Abled Hospital, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Dobbs MB, Gurnett CA. Update on clubfoot: etiology and treatment. Clin Orthop Relat Res. 2009 May;467(5):1146-53. doi: 10.1007/s11999-009-0734-9. Epub 2009 Feb 18. PMID 19224303
- [Background] Engell V, Nielsen J, Damborg F, Kyvik KO, Thomsen K, Pedersen NW, Andersen M, Overgaard S. Heritability of clubfoot: a twin study. J Child Orthop. 2014 Feb;8(1):37-41. doi: 10.1007/s11832-014-0562-7. Epub 2014 Feb 7. PMID 24504418
- [Background] Cady R, Hennessey TA, Schwend RM. Diagnosis and Treatment of Idiopathic Congenital Clubfoot. Pediatrics. 2022 Feb 1;149(2):e2021055555. doi: 10.1542/peds.2021-055555. PMID 35104362
- [Background] Carroll NC. Clubfoot in the twentieth century: where we were and where we may be going in the twenty-first century. J Pediatr Orthop B. 2012 Jan;21(1):1-6. doi: 10.1097/BPB.0b013e32834a99f2. PMID 21946867
- [Background] Owen RM, Capper B, Lavy C. Clubfoot treatment in 2015: a global perspective. BMJ Glob Health. 2018 Sep 3;3(4):e000852. doi: 10.1136/bmjgh-2018-000852. eCollection 2018. PMID 30233830
- [Background] Cooke SJ, Balain B, Kerin CC, Kiely NTJCO. Clubfoot. 2008;22(2):139-49
- [Background] Mejabi J, Esan O, Adegbehingbe O, Orimolade E, Asuquo J, Badmus H, et al. The Pirani scoring system is effective in assessing severity and monitoring treatment of clubfeet in children. 2016;17(4):1-9.
- [Background] Khan MA, Chinoy MA, Moosa R, Ahmed SK. Significance Of Pirani Score at Bracing-Implications for Recognizing A Corrected Clubfoot. Iowa Orthop J. 2017;37:151-156. PMID 28852350
- [Background] Ganesan B, Luximon A, Al-Jumaily A, Balasankar SK, Naik GR. Ponseti method in the management of clubfoot under 2 years of age: A systematic review. PLoS One. 2017 Jun 20;12(6):e0178299. doi: 10.1371/journal.pone.0178299. eCollection 2017. PMID 28632733
- [Background] Verma A, Mehtani A, Sural S, Maini L, Gautam VK, Basran SS, Arora S. Management of idiopathic clubfoot in toddlers by Ponseti's method. J Pediatr Orthop B. 2012 Jan;21(1):79-84. doi: 10.1097/BPB.0b013e328347a329. PMID 21666506
- [Background] Hu W, Ke B, Niansu X, Li S, Li C, Lai X, Huang X. Factors associated with the relapse in Ponseti treated congenital clubfoot. BMC Musculoskelet Disord. 2022 Jan 26;23(1):88. doi: 10.1186/s12891-022-05039-9. PMID 35081931
- [Background] Jowett CR, Morcuende JA, Ramachandran M. Management of congenital talipes equinovarus using the Ponseti method: a systematic review. J Bone Joint Surg Br. 2011 Sep;93(9):1160-4. doi: 10.1302/0301-620X.93B9.26947. PMID 21911524
- [Background] Ponseti IV, Zhivkov M, Davis N, Sinclair M, Dobbs MB, Morcuende JA. Treatment of the complex idiopathic clubfoot. Clin Orthop Relat Res. 2006 Oct;451:171-6. doi: 10.1097/01.blo.0000224062.39990.48. PMID 16788408